CLINICAL TRIAL: NCT02707094
Title: A Pilot Study Examining the Efficacy of Biomodulator Treatment for Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Ann Marie Nayback-Beebe, PhD, RN, COL, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TSNRP-N12-006
Record Dates: First submitted 2014-01-22; First posted 2016-03-14 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Chronic Low Back Pain
Keywords: back; pain; chronic
MeSH Terms: conditions — Pain; Bronchiolitis Obliterans Syndrome | interventions — Immunotherapy; Analgesia; Dosage Forms; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (Medication + Exercise) (Other): Usual Care: Participants will receive guidance on over-the-counter and prescribed pain medications to use to treat their chronic low back pain symptoms. The Research Coordinator (RC) will provide instructions for low back pain stretching and strengthening exercises. The Licensed Provider (LP) will determine if any exercises should be excluded based on their physical limitations. Participants enrolled in the usual care treatment arm will track the frequency of their back stretching and strengthening exercise sessions on the Pain Medication & Exercise Diary. For the purpose of this study, treatment compliance will be met if participants complete the exercises a minimum of three times per week.
  Interventions: Other: Usual Care (Medication + Exercise)
- Biomodulator + Usual Care (Experimental): Biomodulator + Usual Care treatment group: Usual care, as described above, will be provided to all participants randomly allocated to this treatment group, in addition to treatment with the Biomodulator three times per week x 4 weeks. The licensed provider will review medication and treatment logs, prescribe pain medications as indicated, and assess for treatment side effects. In addition to treatment with the Biomodulator, the participant will perform back stretching and core strengthening exercises for a minimum of three times per week as instructed and will be told to use their prescribed pain medications as needed to self-treat their low back pain symptoms (as previously described above).
  Interventions: Device: Biomodulator; Other: Usual Care (Medication + Exercise)

INTERVENTIONS:
Device: Biomodulator — The Biomodulator is a type of very low frequency TENS known as pulsed electromagnetic field therapy (PEMF). Unlike TENS devices that deliver 1-80 milliamperes of electrical current, PEMF devices deliver short bursts of electrical microamperes (millionths of an ampere) to injured tissues without producing heat or interfering with nerve or muscle function. Micro-current levels between 20-500 microampere appear to be most effective at relieving pain and inflammation and promoting tissue healing by realigning the natural electrical balance that exists within the cells that has become disrupted due to injury.
  Other Names: Tennant Biomodulator; Transcutaneous electrical nerve stimulator for pain relief
  Arms: Biomodulator + Usual Care
Other: Usual Care (Medication + Exercise) — The study LP will prescribe an analgesic medication regimen based on the participant's needs. These medications may consist of Non-steroidal anti-inflammatory Drugs (NSAIDs) (ibuprofen, naproxen sodium, etc.), muscle relaxants (Flexeril, Robaxin, valium, etc.), non-narcotic analgesic medications (acetaminophen, aspirin, tramadol, etc.), or narcotic medications (Tylenol #3, Percocet, Vicodin, etc.) depending on the severity of their pain and co-morbid conditions. The RC will also provide instructions for LBP stretching and strengthening exercises. The following exercises will be recommended as a daily regimen: the partial curl, cat and camel, pelvic tilt, quadriceps, arm/leg raises,trunk rotation, single knee to chest stretch, standing hamstring stretch, and double knee to chest stretch.

SUMMARY:
The purpose of this study is to determine the efficacy of self treatment with the Biomodulator device to decrease chronic low back pain (LBP) in active duty service members. In addition, the study will track the use of pain medication and the impact of pain on symptoms of anxiety, depression and Post Traumatic Stress Syndrome (PTSD).

ELIGIBILITY:
Inclusion Criteria:

* active duty Service Members (SMs) between the ages of 18 and 62, inclusive
* history of chronic LBP (i.e. intermittent or continuous LBP symptoms present for 3 months or greater prior to entry into the study
* participants must be using narcotic and/or non-narcotic oral analgesic medications to treat their chronic LBP symptoms on a weekly basis
* must be able to speak and read English and understand the study procedures

Exclusion Criteria:

* pacemaker or implanted electronic device
* history of stroke, blood clots, or cardiac arrhythmias
* pregnancy
* no self-reported history of prescription medication abuse or sole-provider contract for prescribed narcotic medications
* open wound over site of chronic pain;
* history of spinal surgery
* participation in a clinical trial for an investigational drug/ treatment within last 30 days
* undergone treatment with TENS, biofeedback, or acupuncture within last 30 days
* prior treatment with the Biomodulator
* LBP "red flags": fever, trauma, progressive motor or sensory deficit, saddle anesthesia
* participation in the study would delay the medical board (MEB) processing of the service member off of active duty status or would delay a return to duty status to their home unit

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Change over time on the Numerical Rating Scale-11 Pain Score (NRS-11) | Week 0, week 5, week 9

SECONDARY OUTCOMES:
Change over time on the Patient Health Questionnaire -9 (PHQ-9) | Week 0, week 5, week 9
Change over time on the Generalized Anxiety Disorder - 7 (GAD-7) | Week 0, week 5, week 9
Change over time on the Posttraumatic Stress Disorder Checklist - Military (PCL-M) at week 5 | Week 0, week 5, week 9
Change over time on the Pittsburgh Sleep Quality Index (PSQI) | Week 0, week 5, week 9
Change over time on the Oswestry Disability Questionnaire (ODQ) | Week 0, week 5, week 9
Change over time on the Quality of Life - Health Survey (SF-12) | Week 0, week 5, week 9
Change over time on the Interpersonal Relationships Inventory Short Form (IPRI-SF) | Week 0, week 5, week 9
2 questions on treatment perception | week 5
  1. Did you feel this treatment intervention was a success or failure (select one)? Complete Success Partial Success Partial Failure Complete Failure Explain why.
  2. Did you find it easy or difficult to adhere to the treatment plan (select one)? Very Easy Somewhat Easy Somewhat Difficult Very Difficult Explain why.
Abbreviated acceptability rating profile - modified (AARP) | week 5
  Acceptability
Change over time on oral consumption of analgesic medications | Week 0, week 5, week 9

CONTACTS AND LOCATIONS:
Overall Officials: Ann Marie Nayback-Beebe, PhD, FNP-BC, Principal Investigator — Brooke Army Medical Center
Locations (1):
- Brooke Army Medical Center, Fort Sam Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No